CLINICAL TRIAL: NCT06349590
Title: A Phase 1/2 Study of Manipulation of the Gut Microbiome by a Standardized Preoperative Diet to Prevent Colorectal Cancer Recurrence and Metastasis Following Surgery (The DIET Trial)
Brief Title: Manipulation of the Gut Microbiome by a Standardized Preoperative Diet to Prevent Colorectal Cancer Recurrence and Metastasis Following Surgery
Acronym: DIET
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB24-0373
Record Dates: First submitted 2024-03-14; First posted 2024-04-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Intervention Participants (Experimental): Subjects will be provided 21 days of standardized plant-based low fat/ high-fiber meals and complete a food diary up until lunch on the day prior to surgery.
  Interventions: Dietary Supplement: High-fiber/low-fat meals

INTERVENTIONS:
Dietary Supplement: High-fiber/low-fat meals — Meals with Low fat/High fiber

SUMMARY:
A single arm, prospective, single center Phase1/2 Dietary intervention trial for subjects diagnosed with colorectal cancer and scheduled for tumor resection more than 21 days from informed consent. Subjects will be provided 21 days of standardized High-fiber/low-fat meals and complete a food diary up until lunch on the day prior to surgery. Blood samples will be collected at baseline and on the day of surgery. Stool samples will be collected throughout the dietary intervention period at specific timepoints, on the day of surgery, and 30 days post-surgery. Tissue from the tumor resection will be isolated for organoid cultures. Subjects will be followed per standard of care for up to 5 years or disease recurrence, whichever comes first. Subject may be treated for their cancer prior to surgery and/or during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed colorectal adenocarcinoma.
* Planned for primary tumor resection at the University of Chicago Medicine ≥21 from date of obtained informed consent. Patients with metastatic disease but undergoing primary site resection are eligible for the study.
* Age ≥18 years.
* Patients <18 years of age, children are excluded from this study, because they have unique nutritional requirements that might not be met by with the standardized diet. The food in the diet is designed for adults and would not be feasible for children, especially those attending school. In addition, colon cancer is extremely rare in children.
* May have received neoadjuvant therapy (chemotherapy, radiation).
* Patients with Hepatic arterial infusion (HAI) pumps are considered eligible.
* Ability to understand and willing to sign an informed consent, participate in the dietary intervention, collect stools, donate blood, and complete a pre-nutritional evaluation and compliance/patient satisfaction survey.

Exclusion Criteria:

* Previous ostomy (ileostomy or colostomy) or definitive plan for an ostomy (ileostomy or colostomy) during the procedure.
* Antibiotic exposure within 60 days before diet initiation. Antibiotic exposure is defined as a 'course of treatment to treat an infection'. Prophylactic antibiotics prior to a procedure is okay.
* Prebiotic/Probiotic exposure within 60 days before diet initiation.
* Concomitant separate malignancy.
* Allergy to perioperative medications (oral neomycin/metronidazole for bowel preparation, intraoperative prophylactic intravenous cefazolin and metronidazole).
* Patients who are pregnant are not eligible for the study. Pregnant women are excluded from this study because the preoperative diet is not specifically formulated to meet the specific nutritional requirements during the prenatal period.
* History of inflammatory bowel disease
* Severe food allergies precluding the ability to tolerate the standardized dietary intervention.
* Patients with uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Change in lab values of the dietary intervention on the collagenolytic potential of the microenvironment. | At baseline on Day 1 until final values collected on 6 months post-op visit.
  To assess whether the dietary intervention significantly changed the collagenase activity, the site will compare each subject's baseline and final values.

SECONDARY OUTCOMES:
Change in stool samples of the dietary intervention on components of the urokinase-type plasminogen activator (uPA) plasminogen system. | At baseline on Day 1 until final values collected on 6 months post-op visit.
  The site will compare the presence of active-uPA, active- Matrix metalloproteinase-9 (MMP9), and plasminogen in stool samples before and after diet intervention. These assays will be performed in the Shogan Laboratory using western blot and zymography.
Change in stool samples in the metagenomic response of the gut microbiome to the dietary intervention. | At baseline on Day 1 until final values collected on 6 months post-op visit.
  There will be an investigation in the stool associated metagenomics in subjects before and after intervention. During this analysis it will determine the bacterial composition and function, with a particular interest in proteolytic function.
Change in the levels of short-chain fatty acids and bile acids in the metabolomic response to the dietary intervention. | At baseline on Day 1 until final values collected on 6 months post-op visit.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Shogan, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States